CLINICAL TRIAL: NCT05937360
Title: Prevalence of Polycystic Ovary Syndrome In Trinidad
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of The West Indies (Other)
Responsible Party: Principal Investigator, Stephanie Mohammed, Principal Investigator, The University of The West Indies
Other Study IDs: CREC-SA.1723/08/2022
Record Dates: First submitted 2023-06-05; First posted 2023-07-10 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Retrospective Studies

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, buffy coat
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: cross-sectional community based study — Participants (women between the ages of 18 and 45 years) are selected randomly throughout various regions of Trinidad. Every 10th house from the selected regions would be assessed.
  Other Names: retrospective study

SUMMARY:
According to World Health Organization (WHO), in 2010, Polycystic Ovarian Syndrome (PCOS) affected approximately 116 million women worldwide (3.4% of the population). It has been considered one of the most common causes of female infertility and the most common endocrine disorder. The standard diagnosis for the syndrome dates back to international conferences organized by the National Institutes of Health (NIH) in 1990 and the Rotterdam European Society of Human Reproduction and Embryology/ American Society for Reproductive Medicine (ESHRE/ASRM) sponsored PCOS consensus workshop group in 2003 and 2004. Clinical manifestations of the disease may include menstrual irregularities, amenorrhea, ovulation-related infertility, polycystic ovaries, and signs of androgen excess such as acne and hirsutism. This condition may also lead to chronic diseases such as obesity, type 2 diabetes (T2D), dyslipidaemia, and cardiovascular events. Despite the increasing knowledge concerning PCOS, the global picture of the disorder is deficient in a number of geographic regions. Understanding the global prevalence will help to better assess the public health and economic implications of PCOS in Trinidad, allow for improved screening methods, help elucidate the underlying factors and foster improved understanding of the molecular mechanisms in improving the evolutionary process.

DETAILED DESCRIPTION:
Background According to World Health Organization (WHO), in 2010, Polycystic Ovarian Syndrome (PCOS) affected approximately 116 million women worldwide (3.4% of the population). This condition caused symptoms in about 5-10% of women of reproductive age (12 - 45 years). It has been considered one of the most common causes of female infertility and the most common endocrine disorder. The standard diagnosis for the syndrome dates back to international conferences organized by the National Institutes of Health (NIH) in 1990 and the Rotterdam European Society of Human Reproduction and Embryology/ American Society for Reproductive Medicine (ESHRE/ASRM) sponsored PCOS consensus workshop group in 2003 and 2004 (Rotterdam ESHER/ASRM-sponsored PCOS consensus workshop group 2004). Clinical manifestations of the disease may include menstrual irregularities, amenorrhea, ovulation-related infertility, polycystic ovaries, and signs of androgen excess such as acne and hirsutism. This condition may also lead to chronic diseases such as obesity, type 2 diabetes (T2D), dyslipidemia, and cardiovascular events.

Statement of Problem

Despite the increasing knowledge concerning PCOS, the global picture of the disorder is deficient in a number of geographic regions. Understanding the global prevalence and phenotypic presentation of any common disorder, including PCOS, allows for:

1. A determination of the prevalence and associated morbidities of the disorder, to better assess the public health and economic implications of PCOS in this region.
2. A determination of the phenotype of PCOS in this region, allowing for improved screening methods.
3. The elucidation of underlying environmental or ethnic factors that may affect the prevalence, severity or complications of the disorder, via comparison of data between countries.
4. The elucidation of genetic variants underlying the disorder in this region, fostering and improved understanding of the molecular mechanisms underlying the disorder and a better understanding of the evolutionary selection processes that have paradoxically resulted in the current high prevalence of the disorder in the face of obvious reproductive deficits.

Benefit These data would not only lead to an improved understanding of the public health implications of the disorder in Trinidad but also potentially highlight novel etiologic avenues and therapeutic targets.

Aims and objectives

Primary:

1. To determine the prevalence of PCOS among women of reproductive age (a selected population (18 to 45)) in Trinidad.

   Secondary
2. To determine the distribution of phenotypes among women diagnosed with PCOS in the above objective overall and by ethnicity. PCOS sub-phenotypes are as follows: Phenotype A - clinical and/or biochemical hyperandrogenism (HA) and oligi-/anovulation (OA), and polycystic ovarian morphology (PCOM); B - HA and OA; C - HA and PCOM; and D - OA and PCOM;
3. To determine the risks for, metabolic syndrome, depression, obstructive sleep apnea symptoms, fibroids, and general health issues for PCOS women versus women without PCOS in the age groups 18 - 45 years.
4. To determine the genotype of PCOS in Trinidad. Outcome measures and variables Outcome measures (dependent variables) c) Primary outcome ii) Prevalence of PCOS and its symptoms d) Secondary outcome iv) Phenotype of PCOS v) Genotype of PCOS vi) Prevalence and prevalence rationale for PCOS subphenotypes in Trinidad, odds ratio for metabolic syndrome, depression, obstructive sleep apnea symptoms, fibroids, and general patient health issues, adjusted for age, ethnicity, BMI, treatment (OCP), and socioeconomic parameters.

   Covariates (independent variables)
   1. Socio-demographic variables
   2. Baseline characteristics

   Methodology Study design This is a prospective, cross-sectional study. The study will be conducted among females in Trinidad from different geographical locations.

   Study population Based on a review of nine studies conducted in the general population, a conservative prevalence estimate for PCOS, using the Rotterdam 2003 definition, is 13.4%. Based on this formula, a sample size of 495 untreated individuals will be required to determine the prevalence with an absolute error of 3%. Assuming a 50% enrollment rate, 990 women would need to be approached for study inclusion. The study population will be females of reproductive age from Trinidad.

   Strategies for Sampling, Recruitment and Retention Participants will be samples proportionally from all 8 zones in Trinidad. Approximately 124 women in the reproductive age (18 - 45 years old) will be randomly sampled from each zone. Houses will be numbered and random numbers of these houses will be generated using a random number calculator. In each sampled house, females would be prescreened and those that satisfy our inclusion criteria would be selected.

   Telephone numbers of participants will be obtained and follow-up calls made.

   Sampling units are defined as individual unselected women between the ages of 18 and 45 years, identified in the community. The investigators target power analysis on women who do not use hormonal contraception. The investigators assume a conservative response rate of 50% of sampled women. This response rate includes the following parameters: use of hormone/contraceptive use (15%), excluded due to hysterectomy or ovariectomy (3%), excluded due to pregnancy (2%), refusal to participate (20%), and study drop-out/lost to follow-up (10%).

   A conservative prevalence estimate for PCOS based on a review of nine studies conducted in the general population using the Rotterdam 2003 definition is 13.4%. Using the above formula, a sample size of 495 individuals will be required to determine the prevalence with an absolute error of ±3%. Assuming a 50% enrollment rate, 990 women would need to be approached for study inclusion.

   Selection criteria Inclusion criteria
   1. Female, ages 18 to 45 years., all ethnic backgrounds.
   2. The participants must have at least one of the following two features:

   i) Dermatological signs or complaints of clinical hyperandrogenism such as unwanted facial or body hair, loss of scalp hair (alopecia) or persistent acne (pimple).

   ii) Signs or complaints of ovulatory dysfunction such as irregular menses (oligomenorrhoea, amenorrhea or polymenorrhoea), history of anovulation or ultrasonographic findings of polycystic ovarian morphology.

   Exclusion criteria
   1. Women less than 18 years or older than 45 years
   2. Women who are pregnant at the time of evaluation
   3. Postmenopausal women
   4. Women who had undergone hysterectomy and/or bilateral oophorectomy
   5. Anything that would place the individual at increased risk or preclude the individuals' compliance with or completion of the study.
   6. Unwillingness to participate or difficulty understanding the consent process or the study objectives and requirements.

      Sampling technique A consecutive sampling technique will be used for each phase of the study. Consecutive study participants, who meet the selection criteria and give informed written consent, will be recruited for the study. A unique serial identification number will be given to each study participant until the intended sample is attained.

      Study procedure Potential study participants from selected geographical locations will be invited to participate in the study. A confidential study register containing details of potential study participants (name, age, height, weight, blood pressure and contact phone number) will be kept. Potential study participants will be counseled on the objectives of the study and the study protocol. If the potential participant refuses to participate, no further contact will be made with the participant. Inform consent (see attached) will be obtained from each eligible study participant before recruitment for the study. A subject tracking log for longitudinal observation study will be used to track eligible subjects.

      After an informed consent, data will be collected from each study participant using a standard format in a clinical report form (CRF) for uniform data collection from all participants. Each CRF will contain a unique serial identification number. The CRF will be filled by a suitably trained researcher (including the PI, co-investigators and medically trained research assistants). All CRF will be checked for missing data within 24 hours of completion, and any missing data will be detected and collected immediately.

      Each participant will undergo anthropometric measurements (weight, height, waist, circumference and hip circumference) and physical examination for hirsutism, acne, alopecia, and acanthosis nigricans. Participants with an initial hirsutism (mFG) score of 3 or more will be re-assessed by a physician.

      Laboratory investigations will be scheduled during the morning hours (08:00 to 10:00 hours), for blood collection.

      After overnight fasting (of 8 hours or more), 10 ml of venous blood sample will be collected from each study participant. About half (5 ml) of the venous blood will be collected in an EDTA- containing tube for plasma/DNA and the remaining in a plain tube for serum.

      All blood samples will be stored and transported to the laboratory in cooler boxes containing ice packs immediately after collection. At the laboratory, the sample will be separated into serum, plasma and whole blood by centrifugation for 20 minutes at 3000 rpm. The biological specimens will be stored, in small aliquots (of 0.5 ml), in 1.5 to 2.0 ml plastic containers (about 12 cryovials) able to withstand temperatures of -80 degrees.

      Samples for hormonal assay and initial evaluation will be batched at regular intervals for analysis to provide study participants with timely results, allow classification of participants, and minimize the impact of inter-assay variability. At the end of the study, a repeat analysis of biological samples for androgen levels and insulin estimation will be performed at a reference laboratory (Eric William Medical Science Complex).

      Each subject will also complete the following standardized data instruments or forms as appropriate: FG Score self-assessment, SF-12, and Beck depression inventory assessment (see attached).

      The genetic analysis will be performed at the Laboratory at the Department of Pre-clinical Sciences. The initial evaluation and classification of study participants will be done using the flow chart/diagnostic tree by Prof. Azzizz one of the investigators on this project.

      Related or mimicking disorders will be excluded using history, physical examination, and serum TSH, prolactin and 17-OH progesterone. Participants with hypothyroidism on thyroxine replacement therapy will not be recruited for the study until TSH level is normal. Study participants with elevated 17-OH progesterone 2ng/dl (or 200 ng/dl) will have non-classical congenital adrenal hyperplasia (NCAH).

      Data collection instrument:

      The methods of collecting data for the assessment of study objectives include the use of standardized interview-based medical forms; surveys; physical examinations.

      The CRF developed for this study includes; a clinical and anthropometric section and a laboratory result section. The questionnaire section will seek information on socio-demographic variables, reproductive history with an emphasis on menstrual cycle (dating and regularity) and gynecological history, hirsutism, acne, medications, and family history. The anthropometry and clinical section will document the physical findings such as hirsutism, acne, alopecia, and acanthosis nigricans. Subjects will also complete the following standardized data instruments or forms as appropriate: FG Score self-assessment, SF-12, Beck depression inventory, and Epworth sleepiness scale.

      A summary of initial and follow-up procedures.
      1. Physical Exam

         A physical exam will include:
         * Baseline medical examination and
         * Study specific procedures as outlined above.
      2. Baseline medical examination will include • Waist-to-circumference ratio

         * Height measurement
         * Weight measurement
         * Hirsutism assessment
         * Acne assessment
         * Alopecia assessment
         * Acanthosis nigricans assessment

           * Waist and hip circumferences measurement The following measures will be obtained with the subject standing: a) the waist circumference, measured as the circumferential measurement encompassing the lower borders of the 10th rib at the mid-axillary lines; and b) the iliac crest (hip) circumference, measured as the circumferential measurement obtained at the height of the iliac crests, with the tape maintained parallel to the floor. The waist and hip circumferences will be recorded to the nearest 0.1 cm. The waist divided by the iliac crest (hip) circumference will be used to calculate the waist-hip ratio
           * Hirsutism assessment Hirsutism assessment will be performed using the modified Ferriman-Gallwey (mFG) visual hirsutism score scale, by trained study personnel. Inter-reviewer variation will be assessed between study investigators. Photographic examples of each grade will be provided to investigators, as well as training to study personnel.

      mFG scoring will be performed as follows: • Nine body areas are assessed, including the upper lip, chin, chest, upper back, lower back, upper arm, upper and lower abdomen, and thighs.
      * A score of 0 to 4 is assigned to each area examined, based on the density of terminal hairs. A score of 0 represents the absence of terminal hairs, a score of 1 minimal terminal hair growth, a score of 2 mild terminal hair growth, a score of 3 moderate hair growth, and a score of 4 severe terminal hair growth (i.e., like that of a hairy man).

        o Terminal hairs represent hairs that if not cut or trimmed would grow >5 mm in length, are usually pigmented, and are coarser and harder than the softer surrounding vellus hairs, as they have a compact medulla (core) of melanocytes within.
      * Each body area on the mFG form is circled accordingly, leaving those areas with a score of zero blank.

      The scores are summed up to for the 'Total modified FG score'. If patients use permanent/long term epilation or shave hairs, that fact will be recorded on the mFG score sheet.

      • In addition, all subjects will self-score their body and facial hair growth, marking on the mFG score sheet. The subjects will be provided the same mFG score sheet that is used by medical personnel, and will be instructed by trained personnel to circle on the sheet their own body areas they perceive to be affected by excess hair growth. Before they do so the trained personnel will provide them with a short instructional - covering how mFG is performed, what the scores 0 through 4 mean, what terminal hair growth means, and what each body area covers.

      - Acne assessment Assessment of acne will be made by trained personnel; using a standard acne lesion assessment.

      • Acne is scored according to whether it is grade 1 (mild), 2 (moderate), or 3 (severe). Mild acne is characterized by the presence of few to several papules and pustules, but no nodules.

      • Moderate acne by the presence of several to many papules and pustules, along with a few to several nodules.

      • Severe acne by the presence of numerous or extensive papules and pustules, as well as many nodules.
      * Alopecia assessment The Ludwig Scale will be used to diagnose the severity of female hair loss. From left to right in the image below, these Types include Class I, Class II, and Class III: (Attached)
      * Acanthosis nigricans assessment

        * All areas demonstrating acanthosis nigricans should be checked and indicated (see attached).
        * No score is used to denote severity.

3. Screening blood samples for evaluation PCOS Inclusion/Exclusion labs

* TSH**
* PRL**
* 17-OHP***
* P4++
* oGTT** * To be determined in the local clinical lab (MDS Biochemistry Laboratory) in UWI, Trinidad.

  * All subjects. *** For subjects with oligomenorrhea and/or hirsutism and/or PCOM only, who do not use Hormonal Contraception (HC).

    * For subjects with hirsutism and/or PCOM, who have apparently regular menstrual bleeding a day 22-24 progesterone (P4) level will be obtained.

FUNCTIONAL TESTING Adrenocorticotropic Hormone (ACTH) Stimulation Test

An acute ACTH stimulation test is a clinical test performed to exclude 21-hydroxylase deficient nonclassic congenital adrenal hyperplasia (NC-CAH), if the screening (basal) 17-hydroxyprogesterone (17-HP) level is 2 ng/mL (200 ng/dL) or 6.0 nmol/L. This test may also be performed on included subjects, such as controls, for further phenotyping. For androgen excess and/or PCOS patients, an ACTH stimulation test may be part of their standard clinical evaluation if basal 17-HP levels are elevated. The test will be performed as follows:

* The subject will come in between 7-10 am in the morning.
* A small indwelling catheter will be placed in a vein in an arm and a blood sample is drawn through the intravenous catheter (0 min sample).
* 250 mcg of 1-24 ACTH (Cortrosyn®) is then injected through the catheter. The injection is performed over 60 seconds by a physician.
* Sixty minutes after the injection, a second blood sample (60 min, sample) is drawn. • The total amount of blood drawn is 60 ml.

Laboratory evaluations and sample storage in research. Research lab

* SHBG
* Total and Free Testosterone
* DHEAS
* Blood for DNA extraction for later genetic analysis • Extra blood for repository

DNA Core Facility The investigators will obtain blood for DNA extraction since all subjects will undergo standard phenotyping. Blood (in EDTA tubes) will be sent to the Biochemistry Laboratory at Preclinical Sciences, UWI where DNA will be extracted and stored for future analyses. The primary purpose is to serve as a repository to participate in genome wide association studies. In both cases, there will be no release of personal identifiers, and we the investigaotrs will obtain a Certificate of Confidentiality, as done in prior studies. This will be a part of the initial protocol, though subjects will have the option to opt out of this segment of the study or limit the use of their specimen on the consent form. This resource may also prove useful for genome wide association studies or other studies of the genetics of PCOS, oligomenorrhea, and hyperandrogenism.

At this time no genetic analyses are proposed as the number of subjects being collected are insufficient for any significant genetic study. However, as it is the investigators hope that this study will serve as the anchor for subsequent investigations of women's health and PCOS in Trinidad, the investigators intend to isolate and store DNA in the subjects examined in the study. The samples will be stored at The University of the West Indies. If in the future a decision is made to study the DNA samples accumulated, perhaps along with other samples collected, then we the investigators will apply for an amendment for genetic analysis.

Definitions

Ovulatory dysfunction is defined by:

1. Menstrual dysfunction (MD)

   1. Oligi/amenorrhoea: menstrual interval > 35 days or < 10 cycles per year
   2. Polymenorrhoea: menstrual interval < 26 days
   3. Irregular cycle: menstrual interval > 4 days variation
2. Luteal phase (day 21-24) progesterone

   a. Oligi-ovulation: progesterone level < 4ng/ml
3. Polycystic ovarian morphology (PCOM)

   1. Antral follicular count (AFC) of 12 or more follicles measuring 2-9 mm in at least one ovary.
   2. Ovarian volume 0 cm3 in at least one ovary Clinical hyperandrogenism will be diagnosed using hirsutism defined by modified Ferriman-Gallwey (mFG) score of 6 regardless of the presence or absence or acne and alopecia.

Hyperandrogenemia will be defined as a total testosterone, and/or free testosterone, and androstenedione, and/or DHEAS level above the upper 95th percentile of 100 healthy, non-hirsute eumenorrheic women.

Hyperinsulinemia will be defined as a fasting insulin level above the upper 95th percentile of 100 healthy, non-obese women with normal glucose tolerance and no diabetic history or medication use.

Classifications/Phenotypes:

1. Phenotyping: For further evaluation, participants will be divided by presenting phenotype:

   1. Phenotype 'NOT PCOS' i. On medical history a. Long-term predictable regular monthly menstrual bleeding and b. No chronic endocrine disorder or untreated thyroid disorder; and ii. On physical exam: no evidence of hirsutism (i.e. mFG < 3) iii. On transvaginal ultrasonography (TV-U/S): no evidence of ovarian abnormality and no other clinical abnormality.
   2. POSSIBLE PCOS: subdivide into 7 clinical phenotypes i. Phenotype 'POSS. PCOS-MD only':

   <!-- -->

   1. On medical history: menstrual dysfunction (MD);
   2. On physical exam: no evidence of hirsutism (HIR: i.e. mFG 3); and
   3. On TV-U/S: no PCOM. ii. Phenotype 'POSS. PCOS-MD + PCOM':

   <!-- -->

   1. On medical history: menstrual dysfunction (MD);
   2. On physical exam: no evidence of hirsutism (HIR: i.e. mFG 3); and
   3. On TV-U/S: has PCOM. iii. Phenotype ' POSS. PCOS-HIR only':

   <!-- -->

   1. On medical history: long-term predictable regular monthly menstrual bleeding;
   2. On physical exam: evidence of hirsutism (HIR: i.e. mFG 3); and
   3. On TV-U/S: no PCOM. iv. Phenotype 'POSS. PCOS-PCOM only':

   <!-- -->

   1. On medical history: long-term predictable regular monthly menstrual bleeding;
   2. On physical exam: no evidence of hirsutism (HIR: i.e. mFG 3); and
   3. On TV-U/S: has PCOM.

   v. Phenotype 'POSS. PCOS-MD+HR':
   1. On medical history: menstrual dysfunction (MD);
   2. On physical exam: evidence of hirsutism (HIR: i.e. mFG 3); and
   3. On TV-U/S: no PCOM. vi. Phenotype 'POSS. PCOS - MD+HIR+PCOM':

   <!-- -->

   1. On medical history: menstrual dysfunction (MD);
   2. On physical exam: evidence of hirsutism (HIR: i.e. mFG 3); and
   3. On TV-U/S: has PCOM. vii. Phenotype 'POSS. PCOS - HIR+PCOM':

   <!-- -->

   1. On medical history: long-term predictable regular monthly menstrual bleeding;
   2. On physical exam: evidence of hirsutism (HIR: i.e. mFG 3); and
   3. On TV-U/S: has PCOM.
2. Biochemical Phenotyping: For final evaluation, participants will be divided into 3 major phenotypes:

   1. Hyperandrogenic hyperinsulinemia
   2. Hyperandrogenic, non-hyperinsulinemia, and
   3. Non-hyperandrogenic, non-hyperinsulinemia.

Study Specific Biospecimens

The study staff will store the specimens with the following specifications:

* According to the temperature requirements
* Maintain a written and electronic log of sample receipt
* Maintain an electronic log of sample location
* Maintain a written and electronic log of equipment temperatures (temperatures or conditions will be measured daily at the same time)
* Ensure that the freezers or refrigerators have adequate temperature controls
* Ensure quality assurance of equipment, which includes records of regular maintenance and quality evaluations
* Place the sample in a clearly identified location in the freezer or refrigerator (i.e., bar coded container) • Log the sample/s into a database with the location of sample for easy retrieval.

Reporting Procedures The current study provides minimum to modest additional patient risk than standard of care. All SAEs throughout study participation from the start of the study will be reported within 24 hours (or 1 business day) of learning of the event to the local IRB. Reporting will be accomplished by completing the Serious Adverse Event Report. Only study number will identify subject and no other identifying information will be included on the form. The investigators will include the following information when reporting an adverse event, or any other incident, experience, or outcome as an unanticipated problem to the IRB.

Statistical analysis will be done using SPSS.

Data management and Statistical analysis:

Data entry, data processing, and statistical analysis will be done using IBM Statistical Software for Social Sciences (SPSS, Inc., Chicago, IL) version 20.0. Continuous variables (such as age, anthropometric measurements, laboratory values of assay) will be checked for normality using one-sample Kolmogorov-Smirnoff test, and expressed as means ± standard deviation or median ± interquartile range (for data that are not normally distributed).

Categorical variables (such as race, and socioeconomic characteristics) will be expressed as frequencies with accompanying percentages. Differences between groups will be compared using Pearson's Chi-square test or Fisher's exact test for categorical variables. Odds ratio and the corresponding 95% confidence intervals (CI) will be presented. The student t test and ANOVA will be used to compare differences between groups for normally distributed continuous variables. Comparison of continuous variables that were not normally distributed will be done using a non-parametric (Mann-Whitney U test or Kruskal-Wallis test) inferential statistical test.

Linear and logistic regression analysis (univariate and multivariate) will be performed to evaluate the relationship between dependent and independent variables. Test of statistical significance will be set at a p-value less than 0.05.

Ethical considerations:

This study will be conducted according to the ethical guidelines and principles of The International Declaration of Helsinki, the Guidelines for Good Clinical Practice and the National Code of Health Research Ethics (NCHRE). The Ethical Committee for The University of the West Indies will issue approval. All researchers involved in this research project have received training in the Responsible Conduct of Research.

No participant recruitment will commence until approval is received. Written informed consent will be obtained from all participants before recruitment.

Confidentiality of data:

All information about the participants will be obtained using anonymous questionnaires and shall be kept strictly confidential. The participants will be assured that their identity will be kept in confidence by the investigators and that the results obtained will be presented in aggregate manner.

Beneficence to participants:

No participant in this study will be made to pay for any of the procedures. All study participants with abnormal findings will be notified of the results of their evaluation, and those with abnormal physical, historical, or biochemical findings will be encouraged to undergo further investigation or treatment.

Non-Maleficence to the participants:

All precautions will be taken to reduce the discomfort that may result from the venipuncture.

ELIGIBILITY:
Inclusion Criteria:

1. Female, ages 18 to 45 years., all ethnic backgrounds.
2. The participants must have at least one of the following two features:

i) Dermatological signs or complains of clinical hyperandrogenism such as unwanted facial or body hair, loss of scalp hair (alopecia) or persistence acne (pimple).

ii) Signs or complains of ovulatory dysfunction such as irregular menses (oligomenorrhoea, amenorrhea or polymenorrhoea), history of anovulation or ultrasonographic findings of polycystic ovarian morphology.

Exclusion Criteria:

1. Women less than 18 years or older than 45 years
2. Women who are pregnant at the time of evaluation
3. Postmenopausal women
4. Women who had undergone hysterectomy and/or bilateral oophorectomy
5. Anything that would place the individual at increased risk or preclude the individuals compliance with or completion of the study.
6. Unwillingness to participate or difficulty understanding the consent process or the study objectives and requirements.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Female, ages 18 to 45 years., all ethnic backgrounds.
Study Population: Female, ages 18 to 45 years., all ethnic backgrounds
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of PCOS and its symptoms | 1 year
  To determine the prevalence of PCOS in Trinidad, data collection will include blood collection to assess hormones, thyroids, AMH, IR and other parameters as listed in the procedure. Additionally, participants will be issued a questionnaire (see attached) to assess their demographics, history of medical conditions, sexual activity, medications, contraceptive methods, Menes history, weight, height, waist to hip ratio, physical check for hirsutism and acanthosis will be checked for using various approved scales as provided in the questionnaire.
  The hyperandrogenic features will be evaluated using the modified Ferriman-Gallwey Hirstism Score. Mental health will be assessed using BECKS inventory. Physical activity would be assessed using SF-12 scale. Menstrual irregularities will be assessed using the Ruta Menorrghia Scale

CONTACTS AND LOCATIONS:
Locations (1):
- The University of the West Indies, Saint Augustine, Trinidad and Tobago

IPD SHARING:
Plan to Share IPD: Yes
No identifiers will be used. All participants' information are coded and will continue to be coded and stored on a password-protected computer. The information exclusion of identifiers will be published.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 years

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT05937360/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-29): https://cdn.clinicaltrials.gov/large-docs/60/NCT05937360/ICF_001.pdf